CLINICAL TRIAL: NCT02965131
Title: The Effects of the Anhepatic Phase Extended by Temporary Portocaval Shunt on Anesthetic Sensitivity to Desflurane Administered at Constant Minimum Alveolar Concentration and Its Associative Postoperative Cognitive Function
Brief Title: The Effects of the Anhepatic Phase Extended by Temporary Portocaval Shunt on Anesthetic Sensitivity and Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daegu Catholic University Medical Center (Other)
Responsible Party: Principal Investigator, JongHae Kim, Associate Professor, Daegu Catholic University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CR-16-159
Record Dates: First submitted 2016-11-11; First posted 2016-11-16 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Liver Cirrhoses

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-temporary portocaval shunt (No Intervention): No temporary portacaval shunt is created. Full mobilization of the liver was followed by dissection of the hilar structure.
- Temporary portocaval shunt (Experimental): Temporary portocaval shunt is created when inadvertent massive perihepatic bleeding or technical difficulties due to untypical patients' perihepatic anatomy are encountered during total hepatectomy. Hilar dissection preceded the dissection of the retrohepatic vena cava from the native liver. Its creating prolongs the duration of the anhepatic phase.
  Interventions: Procedure: Temporary portocaval shunt

INTERVENTIONS:
Procedure: Temporary portocaval shunt — The hepatic artery, bile duct, and portal vein are dissected and clamped. The retrohepatic vena cava is preserved with selective clamping of the hepatic veins during total hepatectomy. Then, temporary portocaval shunt is constructed by end-to-end anastomosis of the portal vein stump to the middle and left hepatic vein trunk or by end-to-side anastomosis of the stump to the infrahepatic vena cava depending on the remaining length of the vessels.
  Arms: Temporary portocaval shunt

SUMMARY:
This study aims to investigate the effects of the anhepatic phase extended by temporary portocaval shunt on the sensitivity to desflurane administered at 0.6 age-adjusted minimum alveolar concentration and its associative postoperative cognitive function.

DETAILED DESCRIPTION:
The primary end point of this study is the mini-mental state examination in the Korean version of the consortium to establish a registry for Alzheimer's disease assessment packet (MMSE-KC) score obtained 7 days after living donor liver transplantation (LDLT). A sample size of 78 patients was calculated to detect a difference of 2.5 in the MMSE-KC score 7 days after LDLT between the temporary portocaval shunt (TPCS) and non-TPCS groups, achieving a statistical power of 80% at a two-tailed alpha error of 5% under a standard deviation of 3, an unequal allocation ratio between the groups (non-TPCS:TPCS = 83:33), which is the ratio of both types of surgery performed between May 2011 and October 2013 in our institution, and a drop-out rate of 20%, on the assumption that the Mann-Whitney U test would be performed due to the non-normal distribution of MMSE-KC scores in the TPCS group. A small number of patients was expected to be assigned to the TPCS group based on the number of previous cases in our institution and the stringent exclusion criteria.

The data are presented as the means ± standard deviations for normally distributed data, medians (1st quartile - 3rd quartile) for non-normally distributed data, and numbers of patients (percentage) for qualitative data. The assumption of normality is tested using the Kolmogorov-Smirnov and Shapiro-Wilk tests. If at least one null hypothesis of the two tests is not rejected, the data are determined to be normally distributed. Univariate comparisons between the two groups are performed using independent samples Student's t-test for normally distributed variables, the Mann-Whitney U test for non-normally distributed variables, and Fisher's exact test for categorical variables. If Student's t-test is used, the 95% confidence interval of the mean difference and the corresponding P-value is presented. Repeated measures analysis of variance with post hoc paired Student's t-test using Bonferroni correction is performed for normally distributed variables to determine the significance of between- and within-groups effects and interaction between the variables (group versus phase). To determine the significant interval change in non-normally distributed variables during surgery, Friedman's test with post hoc Wilcoxon signed-rank test under Bonferroni correction is used. For the comparison of within-group changes in the total sum scores and subscores of the MMSE-KC, Wilcoxon signed rank test is used. Rank analysis of covariance is used to compare the MMSE-KC score obtained 7 days after surgery between the groups by controlling for the covariates that are found to correlate with the score based on nonparametric Spearman's correlation analysis. The statistical analysis is performed using IBM SPSS Statistics software, version 19.0.0 (IBM Corp., Armonk, NY, United States). A two-tailed P < 0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis regardless of the concurrent presence of hepatocellular carcinoma

Exclusion Criteria:

* Alcoholic liver cirrhosis
* Acute liver failure
* A history of central nervous system disease (e.g., hepatic encephalopathy)
* Use of psychoactive drugs or alcohol within 6 months before the study
* Flapping tremor affecting handwriting performance necessary for assessing constructional praxis
* Difficulty in communicating with medical personnel
* Bispectral index values more than 60 under the predetermined end-tidal minimum alveolar concentration of desflurane during general anesthesia
* Reoperations
* Failure to wean from mechanical ventilation within 24 hours of arrival in the surgical intensive care unit
* Patient refusal

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2014-02; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Mini-Mental State Examination in the Korean Version of the Consortium to Establish a Registry for Alzheimer's Assessment Packet score | Seven day after living donor liver transplantation

SECONDARY OUTCOMES:
Bispectral index values | During the preanhepatic, anhepatic, and neohepatic

IPD SHARING:
Plan to Share IPD: No